CLINICAL TRIAL: NCT03057145
Title: Phase 1 Combination Study of Prexasertib (LY2606368), CHK1 Inhibitor, and Olaparib, PARP Inhibitor, in Patients With Advanced Solid Tumors
Brief Title: Combination Study of Prexasertib and Olaparib in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geoffrey Shapiro, MD, PhD (Other)
Collaborators: Eli Lilly and Company (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Geoffrey Shapiro, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-573
Record Dates: First submitted 2017-02-10; First posted 2017-02-17 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Solid Tumor
Keywords: Solid Tumor
MeSH Terms: interventions — prexasertib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prexasertib Combine with Olaparib (Experimental): * Olaparib will be administered orally on an intermittent schedule during each 28-day cycle. Exact administration schedule will depend on assigned dose level.
  * Prexasertib will be administered intravenously on Days 1 and 15 of a cycle
  Interventions: Drug: Prexasertib; Drug: Olaparib

INTERVENTIONS:
Drug: Prexasertib — LY2606368 is a checkpoint kinase 1 (CHK1) inhibitor that is being developed as a treatment for patients with advanced cancer
  Other Names: LY2606368
Drug: Olaparib — Olaparib is a poly (ADP-ribose) polymerase (PARP) inhibitor.
  Other Names: Lynparza

SUMMARY:
This research study is studying a combination of targeted therapies as a possible treatment for Advanced Solid Tumors.

The study interventions involved in this study are:

* LY2606368
* Olaparib

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved LY2606368 as a treatment for any disease.

The FDA (the U.S. Food and Drug Administration) has approved Olaparib for ovarian cancer but it has not been approved for other uses.

LY2606368 is a checkpoint kinase 1 (CHK1) inhibitor that is being developed as a treatment for patients with advanced cancer. CHK1 inhibitors work by preventing the cancer cells from being able to repair damaged DNA (one of the building blocks of a cell) which then leads to cell death.

Olaparib is a poly (ADP-ribose) polymerase (PARP) inhibitor. PARP is a protein in the body that repairs damage to DNA. In cells that are rapidly growing such as cancer cells, blocking repair of DNA may be of benefit, since it will cause the cell to die.

In this research study, the investigators are combining LY2606368 with Olaparib in the hopes that it will be a safe combination and that the LY2606368 will enhance how the cancer will respond to Olaparib. In previous laboratory studies performed by treating cancer cells with a CHK1 inhibitor and a PARP inhibitor, it was found that the CHK1 inhibitor was successful in increasing efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study-specific procedures not considered part of routine medical care.
* For enrollment to expansion cohort 2, patients must have high-grade serous ovarian or fallopian tube cancer and documentation of BRCA1 or BRCA2 mutation by a CLIA certified lab.
* Patients must have measurable disease by RECIST version 1.1. Measurable disease is defined as at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20mm (≥ 2cm) with conventional techniques or as ≥ 10mm (≥ 1cm) with spiral computed tomography (CT) scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* There are no limits on prior lines of therapy; however, patients must have recovered to eligibility levels from prior toxicity or adverse events as a result of previous treatment prior to entering the study (except alopecia).
* Age ≥18 years, as no dosing or adverse event data are currently available on the use of prexasertib in combination with olaparib in patients < 18 years of age, children are excluded from this study.
* ECOG performance status 0-1. PERFORMANCE STATUS CRITERIA.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥ 1,500/microliters
  * platelets ≥ 100,000/microliters
  * white blood cells (WBC) ≥ 3 x 109/L
  * hemoglobin ≥ 10 g/dL
  * total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤2.5 x institutional ULN or ≤ 5 x institutional ULN in the setting of liver mets
  * creatinine ≤ 1.5X institutional ULN OR
  * creatinine clearance ≥60 mL/min by Cockcroft-Gault equation for participants with creatinine levels above institutional normal.
* The effects of prexasertib and olaparib on the developing human fetus are unknown. For this reason, women of childbearing potential and male patients with partners of childbearing potential must agree to use two highly effective forms of contraception (see Section 5.5.2) prior to study entry, for the duration of study participation, and for 3 months after completion of study. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 3 months after completion of prexasertib and olaparib administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Women of childbearing potential enrolling on study must have a negative serum pregnancy test prior to registration.
* Childbearing potential is defined as women who are not postmenopausal (defined as amenorrheic for ≥ 12 months following cessation of any exogenous hormonal treatments; LH and FSH levels in the postmenopausal range for women under 50; radiation-induced oophorectomy with last menses > 12 months prior; or chemotherapy-induced menopause with last menses > 12 months prior) or surgically sterile (bilateral oophorectomy or hysterectomy).
* Ability to understand and the willingness to sign a written informed consent document. Patients must be willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* Patients must be able to tolerate oral medications and not have gastrointestinal processes that would preclude absorption of olaparib.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Patients who have received prior PARP inhibitor will not be excluded. Patients who have received prior CHK1 inhibitor will be excluded.
* Participants who have undergone major surgery within 14 days of starting the study treatment, or participants who have not recovered to baseline status from the effects of surgery received more than 14 days prior.
* Patients who are receiving any other investigational agents.
* Patients with known brain metastases or carcinomatous meningitis are excluded from this clinical trial, with the exception of patients with brain metastatic disease that has previously been treated and remained stable on MRI ≥ 2 months prior to enrollment, without steroids or anti-epileptic medications. These patients may be enrolled at the discretion of the Principal Investigator.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to prexasertib or olaparib.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled seizures, myocardial infarction within the past 3 months, superior vena cava syndrome, unstable spinal cord compression (untreated and unstable for at least 28 days prior to study entry), or psychiatric illness/social situations that would limit compliance with study requirements. Additionally, patients with other co-morbid disease or metabolic dysfunction that would render the subject at high risk for treatment complications may be excluded at the discretion of the Principal Investigator in the interest of patient safety.
* The effects of prexasertib and olaparib on the developing human fetus are unknown. For this reason, pregnant women are excluded from this study. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with prexasertib and olaparib, breastfeeding women are also excluded.
* Known HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with prexasertib and olaparib. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Participants with known active Hepatitis B or C.
* Participants who have received a previous allogeneic bone marrow transplant.
* Consistent QTc > 470 msec on more than one screening ECGs. Patients with a history of long QTc syndrome or personal or family history of ventricular arrhythmias will be excluded.
* Participants with involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Participants receiving any medications or substances that are strong or moderate inhibitors or inducers of CYP3A4 are ineligible. Please see Section 5.5.1 for further detail and required washout periods. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Participants with a history of myelodysplastic syndrome or acute myeloid leukemia.
* Participants with evidence of pneumonitis on scans at screening will be excluded due to pulmonary toxicities associated with olaparib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 2 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Dose Limiting Toxicity as assessed by CTCAEv4.0 | 1 month
Pharmacokinetic Sampling - Peak Plasma Concentration (Cmax) | 2 months
Pharmacokinetic Sampling - Area Under the Plasma Concentration versus Time Curve (AUC) | 2 months
Anti-Tumor Effects Of The Combination Of Prexasertib And Olaparib by RECIST 1.1 | 2 months
Phospho-CDK Expression In Tumor Biopsies As A Marker Of Prexasertib Effect And Downstream Marker Of Target Engagement | 1 month
RAD51 Focus Formation and γ-H2AX Expression in tumor biopsies Post-Olaparib And Post-Combination Treatment as a marker of DNA damage | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith G, Alholm Z, Coleman RL, Monk BJ. DNA Damage Repair Inhibitors-Combination Therapies. Cancer J. 2021 Nov-Dec 01;27(6):501-505. doi: 10.1097/PPO.0000000000000561. PMID 34904813